CLINICAL TRIAL: NCT06724146
Title: Safety and Efficacy of Upper Arm Combined Treatment Sofwave and Pure Impact to Strength and Tone Muscles and Improve Lax Skin Appearance
Brief Title: Combined Treatment Sofwave and Pure Impact to Strength and Tone Muscles and Improve Lax Skin Appearance
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sofwave Medical LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sofwave25
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Skin Lax and Muscle Strength
Keywords: Upper arm; skin laxity; muscle tone; muscle strength; muscle firm
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Lax Tissue and Muscles (Experimental)
  Interventions: Device: Sofwave and Pure Impact

INTERVENTIONS:
Device: Sofwave and Pure Impact — The Sofwave System, comprised of an applicator and a console, generates high intensity, non-focused ultrasonic energy which can be delivered percutaneously to tissues.
  Pure Impact is an EMS module. This module is wirelessly connected to and controlled by the SofWave console. It functions independently from the existing ultrasound module. Pure Impact generates electrical impulses, which are delivered through electrodes on the skin in direct proximity to the muscles to be stimulated.
  Other Names: SUPERB

SUMMARY:
Open-label, non-randomized, prospective, multi-center, self-controlled clinical study.

DETAILED DESCRIPTION:
Eligible patients will receive combined treatment on both upper arms, included 1 or 2 SofWave treatments and 4 Pure Impact treatments. At the first session (Visit 1), subjects undergo SofWave treatment, and may undergo Pure Impact treatment also at the same visit. If conducting the two procedures on the same day, Pure Impact shall be applied before SofWave. If the procedures are done in separate visits, schedule the Pure Impact 2-7 days after the SofWave procedure. If the two treatments are conducted on the same day, then the second Pure Impact session will be 7-10 days after; similarly, the third and fourth Pure Impact sessions will be performed 7-10 days apart following the previous session. The last (fourth) Pure Impact treatment may occur on the same day or after the optional second SofWave treatment. If conducting the two procedures on the same day, Pure Impact shall be applied before SofWave. If the procedures are done in separate visits, schedule the SofWave 2-7 days after the fourth Pure Impact procedure.

All patients will return to the clinic for two follow-up visits at 4±1 weeks and at 12±2 weeks post last treatment (FU1 and FU2).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 25 years of age and ≤ 70 years of age.
2. Not pregnant or lactating and must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide) or abstinence.
3. Desire to undergo treatments on upper arms for skin lax and for strength and tone muscles.
4. Subject has clearly visible lax skin on the upper arm, which in the investigator's opinion, may benefit from the treatment.
5. Subject agrees to maintain his/her weight (i.e., within 5% of total body weight) by not making any major changes in their diet or exercise routine during the study.
6. Able and willing to comply with all visits, treatments and evaluations schedules and requirements.
7. Willing to have research photos taken of treatment areas.
8. Subject agrees not to undergo any other upper arm skin lax treatments for a period of 3 months following SofWave and Pure Impact treatments.
9. Able to understand and provide written Informed Consent.

Exclusion Criteria:

1. Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breast feeding.
2. Skin disorders (skin infections or rashes, extensive scarring, psoriasis, open wounds etc.) in the treatment area.
3. Medical disorder that would hinder the wound healing or immune response (such as blood disorder) including but not limited to arterial circulation disorders in lower limbs, inflammatory disease, etc.
4. Known allergy to lidocaine or epinephrine.
5. Active malignancy or history of malignancy in the past 5 years.
6. Suffering from significant concurrent illness, such as cardiac disorders, sensory disturbances, diabetes (type I or II), epilepsy, lupus, porphyria, pertinent neurological disorders, uncontrolled hypertension, or liver or kidney disease (i.e. any disease state that in the opinion of the investigator may interfere with the anesthesia, treatment, or healing process).
7. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
8. Suffering from hormonal imbalance, whether related to thyroid, pituitary, or androgen.
9. History of significant lymphatic drainage problems.
10. Currently a heavy smoker or has history of heavy smoking (25 cigarettes per day or more) in past 10 years.
11. History of chronic drug or alcohol abuse.
12. History of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
13. BMI>30kg/m2
14. Non-stable weight nominally ±5% in the past month.
15. Active implanted device such as a pacemaker, defibrillator, drug delivery system or any other metallic or electric implant anywhere in the body.
16. Permanent implant in the treated area such as metal plates, screws and metal piercing, silicone implants or an injected chemical substance, unless deep enough in the periosteal plane.
17. History of epidermal or dermal disorders (particularly involving collagen or microvascularity), including collagen vascular disease or vasculitic disorders.
18. History of a fat reduction procedure (e.g., liposuction, surgery, lipolytic agents, etc.).
19. History of prior surgery in the upper arms.
20. Excessive subcutaneous fat on the upper arms.
21. Severe solar elastosis on the intended to treat area.
22. Significant scarring, atrophic scars in the area to be treated, or has a history of atrophic scars or keloids or prone to bruising.
23. Tattoo or former tattoo at or near treatment area.
24. Muscle atrophy.
25. Need for muscle rehabilitation.
26. Persistent pain at the treated area.
27. Any sensitivity for hydrogel (Pure Impact electrodes pads are made of hydrogel).
28. History of ablative or non-ablative resurfacing/rejuvenation laser treatment or light treatment within the past 6 months, dermabrasion or deep peeling within the past 12 months on the intended to treat area.
29. Inability to understand the protocol or to give informed consent.
30. Unable or unwilling to comply with the study requirements and procedures.
31. Currently enrolled in a clinical study of any other unapproved investigational drug or device.
32. Any other condition that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in the appearance of lax skin | 3 months post treatment follow-up visit
  Rate of improvement in the appearance of lax skin and in the strength and tone muscles in the upper arms following Sofwave and Pure Impact combined treatment based on Global Aesthetic Improvement Scale, as evaluated by independent masked reviewers.

CONTACTS AND LOCATIONS:
Locations (1):
- Tennessee Clinical Research Center, Nashville, Tennessee, United States